CLINICAL TRIAL: NCT00940784
Title: MPD-RC 108: Phase II, Randomized, Double-Blind, Placebo Controlled International Study of Clopidogrel and Aspirin for the Treatment of Polycythemia Vera
Brief Title: Clopidogrel and Aspirin for the Treatment of Polycythemia Vera
Acronym: ISCLAP
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Could not get drug
Sponsor: Ronald Hoffman (Other)
Collaborators: Myeloproliferative Disorders-Research Consortium (Network); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Ronald Hoffman, Professor of Medicine, Hematology and Medical Oncology, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 07-0548-00108; P01CA108671-01A2 (NIH); MPD-RC 108 (Other: Myeloproliferative Disorders-Research Consortium)
Record Dates: First submitted 2009-07-14; First posted 2009-07-16 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Polycythemia Vera
MeSH Terms: conditions — Polycythemia Vera | interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clopidogrel (Experimental): Subjects will be randomized to clopidogrel (oral-75 mg per day) in addition to low dose aspirin and hydroxyurea
  Interventions: Drug: Clopidogrel (Plavix); Drug: Aspirin
- Placebo (Placebo Comparator): Subjects will be randomized placebo in addition to low dose aspirin and hydroxyurea
  Interventions: Drug: Placebo; Drug: Aspirin

INTERVENTIONS:
Drug: Clopidogrel (Plavix) — Clopidogrel, aspirin plus hydroxyurea 75mg qd (Plavix) + 81 - 100 mg qd (aspirin) + hydroxyurea
  Other Names: Plavix
  Arms: Clopidogrel
Drug: Placebo — Placebo, aspirin (81-100 mg qd) plus hydroxyurea
  Arms: Placebo
Drug: Aspirin — 81-100 mg qd

SUMMARY:
Clopidogrel (Plavix) and aspirin are two antithrombotic agents (blood thinners) commonly used in patients with previous thrombotic events (stroke or heart attack). Thrombosis is the formation of a blood clot in a blood vessel. Patients with polycythemia vera are routinely treated with aspirin which has been shown to be effective in reducing their thrombotic risk. However, in polycythemia vera patients with previous thrombosis, a further benefit might be obtained by using the combination of aspirin and clopidogrel which is routinely used in patients with recent acute myocardial ischemia (reduced blood supply to the heart muscle). The study will assess whether this combination therapy greatly increases the risk of bleeding versus aspirin alone, if clopidogrel reduces biological factors that might lead to a stroke or heart attack, and whether a high number of patients with polycythemia vera are resistant to clopidogrel.

Approximately 200 subjects will be enrolled to the Myeloproliferative Disorders-Research Consortium (MPD-RC) study in Europe and the United States with participation expected to last for 7 months (6 months of receiving study medication plus a 30 day follow-up visit).

ELIGIBILITY:
Inclusion Criteria

Patients are included in the study if all of the following criteria are met:

1. A documented diagnosis of polycythemia vera established within 5 years of registration. There must be documentation that the patient has met the revised WHO criteria for the diagnosis of polycythemia vera. Patients must meet the 2 major criteria and 1 of the minor criteria. To verify that the criteria have been met, the appropriate laboratory or pathology reports must be submitted demonstrating that the patient has documentation of these diagnostic criteria.

   Major Criteria:
   * Hemoglobin >18.5 g/dl in men, >16.5 g/dl in women or other evidence of increased red cell volume.
   * Presence of JAK2V617F or other functionally similar mutation such as JAK2 exon 12 mutation

   Minor Criteria:
   * Bone marrow biopsy showing hypercellularity for age with trilineage growth (panmyelosis) with prominent erythroid, granulocyte, and megakaryocytic proliferation.
   * Serum erythropoietin level below the reference range for normal.
   * Endogenous erythroid colony formation in vitro.
2. High cardiovascular risk due to having experienced a prior vascular event such as an ischemic stroke, myocardial infarction or venous thromboembolism. Objective documentation of these events must be accurately reviewed and registered. Stroke and pulmonary embolism must be documented by an imaging study, deep vein thrombosis by ultrasound or other objective methods, myocardial infarction by typical ECG changes and/or an increase in serum troponin. Minor thrombotic events such as transient ischemic attacks, superficial thrombophlepitis or atypical microcirculatory disturbances alone or in combination are considered to qualifying events.
3. No contraindication to aspirin use such as allergy, a history of a previous hemorrhagic stroke or a major gastrointestinal bleed in the previous three months.
4. Use of hydroxyurea as a cytoreductive agent.
5. Signed informed consent: Patients must have signed consents for both the ISCLAP protocol and for the mandatory correlative biomarker MPD-RC 107 protocol in order to be eligible.
6. Serum bilirubin levels less and or equal to 2 times the upper limit of the normal range for the laboratory (ULN).
7. Serum glutamic-pyruvic transaminase (SGPT) alanine aminotransferase [ALT]) levels and serum aspartate aminotransferase (AST) less and or equal 2 x ULN.
8. Serum creatinine levels less and or equal 1.5 x ULN.
9. Women of childbearing potential must have a negative serum or urine pregnancy test prior to clopidogrel treatment and should be advised to avoid becoming pregnant. Women of childbearing potential must practice effective methods of contraception (those generally accepted as standard of care measures). Women of child bearing potential are women who have not been menopausal for 12 months or who have not undergone previous surgical sterilization. If the subject is a woman of childbearing potential, she must use a medically acceptable form of contraception during the study period and for 30 days thereafter.
10. Age greater than or euql to 18 years to 81 years of age. Exclusion Criteria

Subjects are excluded from participating in this study if 1 or more of the following criteria are met:

1. Therapy with clopidogrel within the last 12 months.
2. Any history of prior treatment with aspirin which has resulted in a significant clinical adverse event requiring the discontinuation of aspirin therapy (e.g. bleeding, GI intolerance, etc. or intolerance to aspirin.
3. Patients requiring anticoagulation treatment with warfarin, heparin or low molecular weight heparin for any medical condition.
4. Nursing and pregnant females. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her physician immediately.
5. History of a major bleeding event (requiring blood transfusion or hospitalization, bleeding at a critical site, or life-threatening).
6. Clinical indication for the use of clopidogrel and/or a different antithrombotic regimen.
7. History of active substance or alcoholic abuse within the last year.
8. Known hypersensitivity or contraindication to study treatments.
9. Chronic viral hepatitis or chronic liver disease from any other cause associated with a MELD score equal to or higher than 8.
10. Presence of any disease (e.g. cancer) that is likely to significantly shorten life expectancy.
11. > 81 years of age
12. New York Heart Association (NYHA) Grade II or greater congestive heart failure.
13. A history of gastrointestinal bleeding in the last 12 months.
14. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days, or anticipation of the need for major surgical procedure during the course of the study.
15. Biopsy or other minor surgical procedure, excluding placement of a vascular access device or bone marrow biopsy, within 7 days prior to study enrollment.
16. Ongoing serious, non-healing wound, ulcer, or bone fracture.
17. Treatment with a CYP3A4 inhibitor, including azole antifungals (topicals are permitted); protease inhibitors; nefazodone; cyclosporine; erythromycin; clarithromycin; and troleandomycin.
18. Serum AST greater than or equal to 2 x ULN Serum ALT greater than or equal 2 x ULN Total Bilirubin greater than or equal 2 X ULN Serum creatinine greater than or equal 1.5 X ULN
19. Patients with a diagnosis of polycythemia vera > 5 years from the time of registration
20. Patients who do not have high risk polycythemia vera as defined by experiencing a thrombotic event (see section 3.1) occurring since the initial diagnosis of PV.

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To determine the safety and efficacy of using Clopidogrel plus aspirin on Polycythemia Vera patients | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Hoffman, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai